CLINICAL TRIAL: NCT07137533
Title: Long-Term Peri-Implant Outcomes of Mandibular Overdentures and All-on-4 Prostheses With PEEK Frameworks
Brief Title: Mandibular Overdentures vs All-on-4 With PEEK
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, Dr, Menoufia University
Other Study IDs: ADMNF-00625
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Bone Loss in Jaw

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A - Overdenture Group: Patients in this group received four parallel implants placed in the interforaminal region-two in the lateral incisor sites and two in the first premolar sites. The implants supported a removable overdenture retained by a CAD/CAM-fabricated PEEK framework. The overdentures were designed for improved retention, stability, and load distribution, with acrylic resin denture teeth.
  Interventions: Other: Mandibular Four-Implant-Retained Overdenture (PEEK Framework); Mandibular All-on-4 Fixed Prosthesis (PEEK Framework)
- Group B - Fixed Prosthesis Group: Patients in this group received four implants according to the All-on-4 protocol-two anterior straight implants in the lateral incisor region and two posterior tilted implants in the first premolar region. The implants supported a screw-retained full-arch fixed prosthesis with a CAD/CAM-fabricated PEEK framework and acrylic resin denture teeth. The design aimed to optimize anteroposterior spread and reduce cantilever length while providing a fixed restoration.
  Interventions: Other: Mandibular Four-Implant-Retained Overdenture (PEEK Framework); Mandibular All-on-4 Fixed Prosthesis (PEEK Framework)

INTERVENTIONS:
Other: Mandibular Four-Implant-Retained Overdenture (PEEK Framework); Mandibular All-on-4 Fixed Prosthesis (PEEK Framework) — Group I: Four-implant-retained mandibular overdenture with a CAD/CAM-milled PEEK framework and acrylic denture teeth, retained via attachment mechanisms; implants placed in lateral incisor and first premolar sites; delayed loading protocol.
  Group II: Mandibular All-on-4 fixed prosthesis with a CAD/CAM-milled PEEK framework and acrylic denture teeth; two anterior straight and two posterior tilted implants placed in lateral incisor and first premolar sites; delayed loading protocol.

SUMMARY:
This study compares long-term peri-implant outcomes between two mandibular full-arch rehabilitation approaches-four-implant-retained overdentures and All-on-4 fixed prostheses-when both are fabricated with polyetheretherketone (PEEK) frameworks. While overdentures and All-on-4 prostheses are widely used, evidence on the clinical performance of PEEK frameworks in these modalities is scarce. By evaluating marginal bone loss and other peri-implant parameters, the research aims to clarify whether prosthetic design influences biological outcomes when using this high-performance polymer.

DETAILED DESCRIPTION:
Mandibular edentulism significantly compromises mastication, speech, and psychosocial well-being. Implant-supported prostheses-particularly four-implant-retained overdentures and the All-on-4 full-arch fixed prosthesis-are well-established solutions for restoring function and quality of life. The overdenture approach provides a removable, cost-effective option with enhanced retention and stability, while the All-on-4 concept offers a fixed, immediately functional solution by placing two anterior straight implants and two posterior tilted implants within the interforaminal region.

Long-term success of both treatment modalities is influenced by peri-implant outcomes, especially marginal bone loss (MBL), which reflects the biological stability of the implant-bone interface. MBL can be affected by multiple factors, including loading protocols, implant angulation, prosthetic design, and material properties of the prosthetic framework.

Recent advances in materials science have introduced polyetheretherketone (PEEK), a high-performance polymer, as a promising alternative to traditional metallic frameworks such as titanium or cobalt-chromium. PEEK offers mechanical properties that closely mimic bone, excellent biocompatibility, chemical stability, and a lower elastic modulus that may provide beneficial shock absorption, potentially reducing stress on implants and peri-implant bone. When fabricated via CAD/CAM technology, PEEK frameworks achieve high marginal accuracy and favorable fracture resistance, while also being lightweight and comfortable for patients.

Despite growing interest in PEEK for dental applications, most clinical research has focused on its use in removable partial dentures or single crowns. Data on its performance in full-arch implant prostheses-whether overdentures or All-on-4 fixed restorations-are scarce. Moreover, few studies have directly compared the peri-implant outcomes of these two rehabilitation strategies when using the same framework material.

ELIGIBILITY:
Inclusion Criteria:

Adults aged ≥40 years.

Completely edentulous mandible for at least 6 months prior to implant placement.

Treated with either:

Four-implant-retained mandibular overdenture with a PEEK framework, or

Mandibular All-on-4 fixed prosthesis with a PEEK framework.

All implants placed in the lateral incisor and first premolar regions (per respective protocol).

Restorations fabricated via CAD/CAM-milled PEEK framework with acrylic denture teeth.

Prosthesis delivered with a delayed loading protocol.

Minimum clinical and radiographic follow-up of 4 years.

Availability of standardized baseline and follow-up periapical radiographs for marginal bone level assessment.

Treated by the same surgical and prosthodontic team.

Exclusion Criteria:

History of uncontrolled systemic diseases that could affect bone healing (e.g., uncontrolled diabetes, osteoporosis under bisphosphonate therapy).

History of head and neck radiotherapy.

Active periodontal or peri-implant infection at the time of implant placement.

Insufficient bone volume in the interforaminal region requiring grafting beyond minor augmentation.

Heavy smoking habit (>10 cigarettes/day) at the time of treatment.

Parafunctional habits (e.g., severe bruxism or clenching) documented in patient records.

Use of medications known to affect bone metabolism (e.g., high-dose corticosteroids, antiresorptive drugs).

Pregnancy at the time of implant placement.

Incomplete clinical or radiographic records.

Follow-up period of less than 4 years.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients with completely edentulous mandibles who underwent full-arch implant-supported rehabilitation between 2015 and 2018 at two private dental clinics. Eligible patients had been restored with either a four-implant-retained mandibular overdenture or an All-on-4 mandibular fixed prosthesis, both fabricated with CAD/CAM-milled polyetheretherketone (PEEK) frameworks and acrylic denture teeth. All implants were placed in the inter foraminal region, following a delayed loading protocol.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss (MBL) per implant (mm) | 5 years
  Definition: Change in crestal bone level on the mesial and distal aspects of each implant from baseline to last follow-up.
  Baseline: Prosthesis delivery (insertion) radiograph.
  Follow-up window: Minimum 48 months post-insertion (target range ≈ 4-9 years, depending on patient record length).
  Measurement method: Standardized periapical radiographs using a paralleling technique

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
Up on resonable request from the corresponding author